CLINICAL TRIAL: NCT02923518
Title: Cardiac Screening of Middle Aged and Older Women and Men (Master Athletes) Who Participate in Long Distance Endurance Training and Competitions.
Brief Title: Cardiac Screening of Middle Aged and Older Women and Men (Master Athletes)
Acronym: MASTERSCREEN
Status: Completed | Type: Observational
Sponsor: LHL Helse (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/21007
Record Dates: First submitted 2016-10-01; First posted 2016-10-04 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Heart Disease
Keywords: Heart Screening; Master Athletes; Cardiovascular Disease
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Inclusion group: Inclusion group: Those with a positive score in a questionnaire including symptoms and family history and/or high risk-score in the NORRISK-score system.
  Interventions: Other: Questionnaire
- Control group: Those without a positive score on the two scores listed above.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Observational study without any intervention described under intervention type

SUMMARY:
In 2010 there was published new European recommendations for assessment of adult and elderly men and women, who want to start with physical activity and/or participate in endurance contests. In this study we want to test if a group of people with positive score on a self-reported questionnaire and/or high-risk score in a risk scoring system (NORRISK) have more undetected heart diseases than a control group with no reported or detected risk factors.

DETAILED DESCRIPTION:
Forty senior athletes between 35 to approximately 80 yrs old with a positive score will be included in one group, and another forty seniors without positive score in a control group. Each of them will be tested with an cardiorespiratory exercise test (CPET) with ECG and examined with echocardiography together with an usual medical examination and blood tests (cholesterol and HbA1c-glucose). Some with symptoms of arrhythmias will be examined by 24-hours Holter-monitoring.

The main purpose of the study is to assess if men and women with a positive score on the questionnaire og NORRISK-screening (risk calculator for coronary heart disease) have more detectable heart diseases than the control group.

ELIGIBILITY:
Inclusion Criteria:

> 35 yrs old Master athletes Positive score on symptom based questionnaire or high risk score No known heart disease Participated in long-term endurance competitions

Exclusion Criteria:

< 35 yrs old Known heart disease

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Senior men and women < 35 yrs participating in long-enurance competitions. 40 persons in a group with positive score and one group without.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2016-10; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Differences among two groups of senior athletes in detecting heart diseases by a screening program | One year
  Examine if a simple screening program is efficient in detecting heart diseases

CONTACTS AND LOCATIONS:
Overall Officials: Hege Lundring, M.D., Study Director — General manager the LHL-clinics
Locations (1):
- LHL-clinics Feiring, Feiring, Norway

IPD SHARING:
Plan to Share IPD: No